CLINICAL TRIAL: NCT03022942
Title: Efficacy of Costal Mobilization Techniques and Diaphragm Release in Thoracoabdominal Kinematics, Diaphragm Mobility and Submaximal Functional Capacity in Patients With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial
Brief Title: Efficacy of Costal Mobilization Techniques and Manual Diaphragm Release Technique in Patients COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, HELENA MEDEIROS ROCHA, Graduate, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Lacap UFPE
Record Dates: First submitted 2016-12-22; First posted 2017-01-18 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Copd; Chest Disorders; Diaphragmatic Disorder
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costal mobilization & Diaphragm Release (Experimental): Costal mobilization. Lying: two sets of ten deep respiratory cycles with one minute interval between sets. Sitting: two series with interval of one minute between them. Manual Diaphragm Release Technique: will be applied during two series of ten deep respiratory cycles, with one minute interval between sets.
  Interventions: Other: GROUP Costal mobilization & Diaphragm Release
- Manual Diaphragm Release (Active Comparator): Manual Diaphragm Release Technique: will be applied during two series of ten deep respiratory cycles, with one minute interval between sets.
  Interventions: Other: GROUP Manual Diaphragm Release

INTERVENTIONS:
Other: GROUP Costal mobilization & Diaphragm Release — Costal mobilization technique (Rib raising): The patient will be lying. The Therapist supports the last four pulps of both hands at the rib angles, gently traverses the rib angles in the posterior-anterior direction, using the stretcher as a lever to facilitate the elevation of the costal angles. Siting: The Therapist hugs the patient by supporting the ribs of the fingers at the rib angles, gently traverses the rib angles bilaterally in the anterior-lateral direction. Manual Diaphragm Release Technique: The therapist makes manual contact with the underside of the costal border of the common cartilage of the last rib. In the inspiratory phase, the therapist draws the points of contact with both hands in a cephalad direction and slightly Accompanying the movement of the rib cage.
  Other Names: GROUP Rib Raising & Diaphragm Release; GROUP A
  Arms: Costal mobilization & Diaphragm Release
Other: GROUP Manual Diaphragm Release — The therapist makes manual contact with the underside of the costal border of the common cartilage of the last rib. In the inspiratory phase, the therapist draws the points of contact with both hands in a cephalad direction and slightly Accompanying the movement of the rib cage.
  Other Names: GROUP B
  Arms: Manual Diaphragm Release

SUMMARY:
To evaluate the acute and chronic effects of costal mobilization techniques and diaphragmatic release in chest cavity kinematics, diaphragmatic mobility and functional capacity in patients with chronic obstructive pulmonary disease

DETAILED DESCRIPTION:
Study will be a controlled clinical trial in which participants will be randomized into 2 groups: GROUP A (costal mobilization techniques and Manual Diaphragm Release Technique), GROUP B (Manual Diaphragm Release Technique). After the initial evaluation, participants will undergo six sessions of care according to randomization and will be reevaluated in 3 following situations: immediately after the first session, at the end of treatment and one week after the last session. The evaluation will be performed through Optoelectronic plethysmography , Pollar, Ultrasound and 6-minutes walk test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (spirometry with FEV1 <80% and FEV1 / FVC <0.7) of both sexes, who are not undergoing another physiotherapeutic treatment, from to 21 years of age, clinically stable without exacerbation in the last 6 weeks.

Exclusion Criteria:

* Patients with rheumatic or orthopedic diseases;
* Deformities / abnormalities in the spine that compromise the mechanics of the respiratory system;
* Rib fracture for less than 1 year;
* Respiratory co-morbidities;
* History of thoracic or abdominal surgery for less than 1 year;
* Osteoporosis and IMC > 30kg / m²

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Mobility of the thoracic cage | Three weeks total: Thirty minutes after the first intervention, after two weeks of intervention and after one week without treatment (follow up)
  Will be measured by optoelectronic plestimography

SECONDARY OUTCOMES:
Diaphragma mobility | Three weeks total: Thirty minutes after the first intervention, after two weeks of intervention and after one week without treatment (follow up)
  Will be measured with ultrasonography
functional capacity | Three weeks total: after two weeks of intervention and after one week without treatment (follow up)
  Will be measured six minute walk test
heart rate variability | 1 day: before and after the intervention
  Will be measured Pollar

CONTACTS AND LOCATIONS:
Overall Officials: HELENA M ROCHA, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No